CLINICAL TRIAL: NCT02934048
Title: Optimal Duration of Antimicrobial Susceptibility Test (AST) Guided Rescue Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016SDU-QILU-16
Record Dates: First submitted 2016-10-09; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Therapeutic Duration; Helicobacter Pylori; Antimicrobial Susceptibility Test; Eradication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 7-day triple regimen (Experimental): Patients in this group received a 7-day triple regimen to eradicate H. pylori. The triple therapy contains proton pump inhibitor (PPI)-clarithromycin plus a susceptible antibiotics will be involved in the study.
  Interventions: Other: 7-day triple regimen guided by AST
- 10-day triple regimen (Experimental): Patients in this group received a 10-day triple regimen to eradicate H. pylori. The triple therapy contains PPI-clarithromycin plus a susceptible antibiotics will be involved in the study.
  Interventions: Other: 10-day triple regimen guided by AST
- 14-day triple regimen (Experimental): Patients in this group received a 14-day triple regimen to eradicate H. pylori. The triple therapy contains PPI-clarithromycin plus a susceptible antibiotics will be involved in the study.
  Interventions: Other: 14-day triple regimen guided by AST

INTERVENTIONS:
Other: 7-day triple regimen guided by AST — Patients in this group will receive a 7-day triple regimen to eradicate H. pylori. The regimen is consist of a PPI and 2 susceptible antibiotics which are determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: 7-day triple regimen
Other: 10-day triple regimen guided by AST — Patients in this group will receive a 10-day triple regimen to eradicate H. pylori. The regimen is consist of a PPI and 2 susceptible antibiotics which are determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: 10-day triple regimen
Other: 14-day triple regimen guided by AST — Patients in this group will receive a 14-day triple regimen to eradicate H. pylori. The regimen is consist of a PPI and 2 susceptible antibiotics which are determined by AST. The susceptibility of amoxicillin, clarithromycin, metronidazole, tinidazole,levofloxacin, furazolidone and tetracycline will be evaluated.
  Arms: 14-day triple regimen

SUMMARY:
Strongly evidence supports that H. pylori eradication is an effective approach to reduce the incidence of those pathologies. However, due to the increasing resistance rates to antibiotics, failures of H. pylori eradication get more and more common. Thus, rescue therapy for persistent H. pylori infection is becoming a grand challenge the investigators have to face.

ELIGIBILITY:
Inclusion Criteria:

* Patients require upper endoscopy owing to persistent H. pylori infection despite one or more treatment attempts.

Exclusion Criteria:

* Age younger than 18 years;
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer;
* Known or suspected allergy to study medications;
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The different rate of H. pylori eradication among 3 different course of treatments (7-day, 10-day and 14-day) guided by AST in intention-to-treat (ITT) analysis. | 9 months
The different rate of H. pylori eradication among 3 different course of treatments (7-day, 10-day and 14-day) guided by AST in per-protocol (PP) analysis. | 9 months

SECONDARY OUTCOMES:
the rate of improving dyspepsia symptoms after H. pylori eradication | 9 months
the rate of adverse events happening | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University